CLINICAL TRIAL: NCT03344458
Title: enliGHten: A Multicenter, Phase 3, Long-Term, Open-Label Trial Investigating Safety and Efficacy of TransCon hGH Administered Once-Weekly in Children With Growth Hormone Deficiency (GHD) Who Have Completed a Prior TransCon hGH Clinical Trial
Brief Title: A Long-Term Trial Investigating Safety and Efficacy of TransCon hGH in Children With Growth Hormone Deficiency Who Have Completed a Prior TransCon hGH Clinical Trial
Acronym: enliGHten
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ascendis Pharma A/S (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TransCon hGH CT-301EXT; 2017-003410-20 (EudraCT Number)
Record Dates: First submitted 2017-11-14; First posted 2017-11-17 (Actual); Results first posted 2024-05-08 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-04

CONDITIONS: Growth Hormone Deficiency, Pediatric; Endocrine System Diseases; Hormone Deficiency; Pituitary Diseases
Keywords: Human Growth Hormone; hGH; GHD; rhGH; Pediatric Growth Hormone Deficiency; Long Acting Growth Hormone; Somatropin; Prodrug; Growth Failure; Growth Hormone Replacement Therapy; Sustained Release Growth Hormone; Growth Hormone Deficiency; TransCon GH
MeSH Terms: conditions — Dwarfism, Pituitary; Endocrine System Diseases; Pituitary Diseases; Failure to Thrive

STUDY DESIGN:
Intervention Model Description: All study participants will receive TransCon hGH
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- TransCon hGH (Experimental): Once weekly subcutaneous injection of TransCon hGH
  Interventions: Drug: TransCon hGH

INTERVENTIONS:
Drug: TransCon hGH — Once weekly subcutaneous injection of TransCon hGH

SUMMARY:
A multicenter, phase 3, long-term extension trial of TransCon hGH administered once-weekly in children with growth hormone deficiency (GHD) who previously participated in a phase 3 TransCon hGH trial. Approximately 300 children (males and females) with GHD will be included. All study participants will receive TransCon hGH. This is a global trial that will be conducted in, but not limited to, the United States, Poland, Bulgaria, Ukraine, Armenia, Russia and Australia.

ELIGIBILITY:
Inclusion Criteria:

1. Children who have completed a prior phase 3 TransCon hGH trial
2. Children who have not permanently discontinued study drug in the prior trial
3. Written, signed, informed consent of the parent or legal guardian of the subject and written assent of the subject as required by the IRB/HREC/IEC

Exclusion Criteria:

1. Poorly-controlled diabetes mellitus (HbA1c ≥ 8.0%) or diabetic complications
2. Evidence of closed epiphyses, defined as bone age > 14.0 years for females or > 16.0 years for males
3. Major medical conditions unless approved by Medical Expert
4. Known hypersensitivity to the components of the trial medication
5. Likely to be non-compliant with respect to trial conduct (in regards to the subject and/or the parent/legal guardian/caregiver)
6. Pregnancy
7. Any other reason that in the opinion of the investigator would prevent the subject from completing participation or following the trial schedule

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 298 (Actual)
Dates: Start 2017-12-19 (Actual); Primary Completion 2023-02-21 (Actual); Study Completion 2023-02-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Beckert, MD, Study Director — Ascendis Pharma A/S; Aimee D Shu, MD, Study Director — Ascendis Pharma, Inc.
Locations (41):
- United States (21):
  - Ascendis Pharma Investigational Site, Birmingham, Alabama
  - Ascendis Pharma Investigational Site, Los Angeles, California
  - Ascendis Pharma Investigational Site, Orange, California
  - Ascendis Pharma Investigational Site, Sacramento, California
  - Ascendis Pharma Investigational Site, Centennial, Colorado
  - Ascendis Pharma Investigational Site, Jacksonville, Florida
  - Ascendis Pharma Investigational Site, Orlando, Florida
  - Ascendis Pharma Investigational Site, Tallahassee, Florida
  - Ascendis Pharma Investigational Site, Saint Paul, Minnesota
  - Ascendis Pharma Investigational Site, Jackson, Mississippi
  - Ascendis Pharma Investigational Site, Lebanon, New Hampshire
  - Ascendis Pharma Investigational Site, Mineola, New York
  - Ascendis Pharma Investigational Site, New York, New York
  - Ascendis Pharma Investigational Site, Cleveland, Ohio
  - Ascendis Pharma Investigational Site, Oklahoma City, Oklahoma
  - Ascendis Pharma Investigational Site, Portland, Oregon
  - Ascendis Pharma Investigational Site, Dallas, Texas
  - Ascendis Pharma Investigational Site, Fort Worth, Texas
  - Ascendis Pharma Investigational Site, Charlottesville, Virginia
  - Ascendis Pharma Investigational Site, Norfolk, Virginia
  - Ascendis Pharma Investigational Site, Tacoma, Washington
- Ascendis Pharma Investigational Site, Yerevan, Armenia
- Ascendis Pharma Investigational Site, Clayton, Victoria, Australia
- Ascendis Pharma Investigational Site, Minsk, Belarus
- Ascendis Pharma Investigational Site, Varna, Bulgaria
- Ascendis Pharma Investigational Site, Tbilisi, Georgia
- Ascendis Pharma Investigational Site, Athens, Greece
- Ascendis Pharma Investigational Site, Auckland, New Zealand
- Poland (2):
  - Ascendis Pharma Investigational Site, Gdansk
  - Ascendis Pharma Investigational Site, Warsaw
- Russia (8):
  - Ascendis Pharma Investigational Site, Izhevsk
  - Ascendis Pharma Investigational Site, Krasnoyarsk
  - Ascendis Pharma Investigational Site, Moscow
  - Ascendis Pharma Investigational Site, Saint Petersburg
  - Ascendis Pharma Investigational Site, Saratov
  - Ascendis Pharma Investigational Site, Ufa
  - Ascendis Pharma Investigational Site, Vologda
  - Ascendis Pharma Investigational Site, Voronezh
- Ukraine (3):
  - Ascendis Pharma Investigational Site, Kharkiv
  - Ascendis Pharma Investigational Site, Kyiv
  - Ascendis Pharma Investigational Site, Odesa

REFERENCES:
- [Result] Maniatis AK, Casella SJ, Nadgir UM, Hofman PL, Saenger P, Chertock ED, Aghajanova EM, Korpal-Szczyrska M, Vlachopapadopoulou E, Malievskiy O, Chaychenko T, Cappa M, Song W, Mao M, Mygind PH, Smith AR, Chessler SD, Komirenko AS, Beckert M, Shu AD, Thornton PS. Safety and Efficacy of Lonapegsomatropin in Children With Growth Hormone Deficiency: enliGHten Trial 2-Year Results. J Clin Endocrinol Metab. 2022 Jun 16;107(7):e2680-e2689. doi: 10.1210/clinem/dgac217. PMID 35428884
- See also: Safety and Efficacy of Lonapegsomatropin in Children With Growth Hormone Deficiency: enliGHten Trial 2-Year Results. — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC9202697/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Overall, 298 subjects entered the extension trial from the parent trials: 103 subjects from the CT-301 Lonapegsomatropin group, 55 subjects from the CT-301 Genotropin group, and 140 subjects from the CT-302 Lonapegsomatropin group.
Pre-assignment Details: Patients who completed a prior phase 3 lonapegsomatropin trial were screened. Patients with poorly controlled diabetes or diabetic complications, or with evidence of closed epiphyses or known hypersensitivity to the trial medication were excluded. All inclusion/exclusion criteria were met during enrollment.
Groups:
- Lonapegsomatropin: Once weekly subcutaneous injection of lonapegsomatropin (TransCon hGH)
Period: Overall Study
Arm/Group | Lonapegsomatropin
Started | 298
Completed | 259
Not Completed | 39
Not completed — Physician Decision | 1
Not completed — Withdrawal by Subject | 16
Not completed — Other reasons | 10
Not completed — Lost to Follow-up | 9
Not completed — Protocol Violation | 3

BASELINE CHARACTERISTICS:
Arm/Group | Lonapegsomatropin
Number analyzed (Participants) | 298
Age, Continuous [Mean (Standard Deviation); unit: years] | 10.27 (3.421)
Age, Customized [Count of Participants; unit: Participants]
  Infants and toddlers (28 days-23 months) | 1
  Children (2-11 years) | 196
  Adolescents (12-17 years) | 101
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 63
  Male | 235
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Race
  Participants
    Asian | 6
    Black or African American | 5
    Native Hawaiian or other Pacific Islander | 2
    White | 270
    Multiple | 3
    Other | 4
    Unknown | 8
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Ethnicity
  Participants
    Hispanic or Latino | 15
    Not Hispanic or Latino | 272
    Not reported | 8
    Unknown | 3
Region of Enrollment [Count of Participants; unit: Participants]
  Armenia | 10
  Greece | 3
  New Zealand | 9
  United States | 174
  Ukraine | 11
  Poland | 8
  Georgia | 10
  Australia | 5
  Belarus | 5
  Bulgaria | 3
  Russia | 50
  Canada | 1
  Turkey | 3
  Italy | 3
  Romania | 3
Tanner Stage [Count of Participants; unit: Participants] — The Tanner scale is a Sexual Maturity Rating classification system used to document the development of secondary sex characteristics of children during puberty. The scale ranges from prepubertal (Stage 1) to adult (Stage 5).
  Participants
    Tanner Stage 1 | 214
    Tanner Stage 2 | 40
    Tanner Stage 3 | 25
    Tanner Stage 4 | 16
    Tanner Stage 5 | 3
Height SDS [Mean (Standard Deviation); unit: Height Standard Deviation Score] — Height Standard Deviation Score (SDS) is the number of standard deviations above or below the mean height for age and sex. A Standard Deviation Score of 0 represents the population mean or average. A negative SDS indicates below average height and a positive SDS indicates above average height.
  Height Standard Deviation Score | -1.564 (0.878)
IGF-1 SDS [Mean (Standard Deviation); unit: IGF-1 Standard Deviation Score] — Insulin-like Growth Factor-1 (IGF-1) Standard Deviation Score (SDS) is the number of standard deviations above or below the mean IGF-1 level for age and sex. A standard deviation score of 0 represents the population mean.
  IGF-1 Standard Deviation Score | 0.515 (1.579)

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Treatment-Emergent Adverse Events [Long-Term Safety and Tolerability]
Description: Long-term safety and tolerability of weekly lonapegsomatropin (TransCon hGH) treatment
Time Frame: Up to Week 208
Measure: Count of Participants; unit: Participants
Arm/Group | Lonapegsomatropin
Number analyzed (Participants) | 298
Participants | 226

2. Secondary Outcome: Annualized Height Velocity by Visit
Description: Annualized height velocity (AHV) by visit with long-term dosing of weekly lonapegsomatropin treatment
Time Frame: Up to Week 208
Population: A rolling baseline was used to ensure the baseline was no more than 52 weeks apart. The rolling baseline was used to calculate the annualized height velocity to ensure there was a one-year gap; from the 15-month (65 weeks) visit onwards, the baseline value used for each successive HV calculation was the patient's height at the visit 52 weeks previously. At each post-baseline visit, n is the number of subjects with non-missing baseline and a specific post-baseline.
Measure: Mean (Standard Deviation); unit: cm/year
Arm/Group | Lonapegsomatropin
Number analyzed (Participants) | 298
cm/year
  Week 13: number analyzed (Participants) | 295
  Week 13 | 8.904 (2.795)
  Week 52: number analyzed (Participants) | 284
  Week 52 | 8.560 (1.801)
  Week 104: number analyzed (Participants) | 255
  Week 104 | 7.854 (1.953)
  Week 156: number analyzed (Participants) | 236
  Week 156 | 7.081 (1.838)
  Week 208: number analyzed (Participants) | 148
  Week 208 | 6.462 (1.868)

3. Secondary Outcome: IGF-1 SDS by Visit
Description: Insulin-like Growth Factor-1 (IGF-1) standard deviation score (SDS) by visit with long-term dosing of weekly lonapegsomatropin treatment at Week 13, Week 52, Week 104, Week 156, and Week 208. IGF-1 SDS is the number of standard deviations above or below the mean IGF-1 level for a child of the same age and sex. The target range for IGF-1 SDS was 0 to +2. An IGF-1 SDS of 0 represents the population mean. If the IGF-1 SDS is < 0, then the negative score indicates an IGF-1 below the mean IGF-1 for a child of the same age and sex. If the IGF-1 SDS is > 0, then the positive score indicates an IGF-1 above the mean IGF-1 for a child of the same age and sex. A positive score of IGF-1 SDS indicates a better outcome.
Time Frame: Up to Week 208
Population: At each post-baseline visit, n is the number of subjects with non-missing baseline and specific post-baseline.
Measure: Mean (Standard Deviation); unit: Standard Deviation Score
Arm/Group | Lonapegsomatropin
Number analyzed (Participants) | 298
Standard Deviation Score
  Week 13: number analyzed (Participants) | 290
  Week 13 | 1.210 (1.400)
  Week 52: number analyzed (Participants) | 282
  Week 52 | 1.355 (1.231)
  Week 104: number analyzed (Participants) | 249
  Week 104 | 1.613 (1.189)
  Week 156: number analyzed (Participants) | 231
  Week 156 | 1.453 (1.125)
  Week 208: number analyzed (Participants) | 142
  Week 208 | 1.597 (1.177)

4. Secondary Outcome: Height SDS - Change From Baseline
Description: Change in Height Standard Deviation Score (SDS) from baseline with long-term dosing of weekly lonapegsomatropin treatment at Week 13, Week 52, Week 104, Week 156, and Week 208. Height SDS is the number of standard deviations above or below the mean height for age and sex. A Standard Deviation Score of 0 equals the population mean. If the Height SDS is < 0, then the negative score indicates a height below the mean height for a child of the same age and sex. If the Height SDS is > 0, then the positive score indicates a height above the mean height for a child of the same age and sex. A positive change from baseline in Height SDS indicates improved outcomes.
Time Frame: Up to Week 208
Population: At each post-baseline visit, n is the number of subjects with non-missing baseline and specific post-baseline.
Measure: Mean (Standard Deviation); unit: Standard Deviation Score
Arm/Group | Lonapegsomatropin
Number analyzed (Participants) | 298
Standard Deviation Score
  Week 13: number analyzed (Participants) | 295
  Week 13 | 0.141 (0.125)
  Week 52: number analyzed (Participants) | 284
  Week 52 | 0.491 (0.307)
  Week 104: number analyzed (Participants) | 255
  Week 104 | 0.841 (0.487)
  Week 156: number analyzed (Participants) | 236
  Week 156 | 1.089 (0.534)
  Week 208: number analyzed (Participants) | 148
  Week 208 | 1.242 (0.652)

ADVERSE EVENTS:
Time Frame: From Informed Consent Form signature up to 14 days after the final dose, up to 260 weeks.
Description: A treatment-emergent adverse event (TEAE) was defined as any adverse event that first occurred or worsened after the first trial drug dose and before the end of the trial. Each subject was counted only once within each preferred term.
Arm/Group | Lonapegsomatropin
All-Cause Mortality (participants affected / at risk) | 0/298
Serious Adverse Events (participants affected / at risk) | 21/298
Other Adverse Events (participants affected / at risk) | 225/298
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lonapegsomatropin (N=298)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1)
Forearm fracture (Injury, poisoning and procedural complications) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1)
Limb injury (Injury, poisoning and procedural complications) | 1 (1)
Lip injury (Injury, poisoning and procedural complications) | 1 (1)
Upper limb fracture (Injury, poisoning and procedural complications) | 1 (1)
Diverticulitis Meckel's (Congenital, familial and genetic disorders) | 1 (1)
Brain stem infarction (Nervous system disorders) | 1 (1)
Epilepsy (Nervous system disorders) | 1 (1)
Generalised tonic-clonic seizure (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Serum sickness-like reaction (Immune system disorders) | 1 (1)
Cyclic vomiting syndrome (Gastrointestinal disorders) | 1 (6)
Inguinal hernia (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Adenoidal hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nephrotic syndrome (Renal and urinary disorders) | 1 (1)
Scoliosis (Musculoskeletal and connective tissue disorders) | 1 (1)
COVID-19 (Infections and infestations) | 3 (3)
Pneumonia (Infections and infestations) | 2 (2)
Abscess (Infections and infestations) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1)
Gastroenteritis salmonella (Infections and infestations) | 1 (1)
Gastrointestinal viral infection (Infections and infestations) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1)
Tonsillitis (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lonapegsomatropin (N=298)
SARS-CoV-2 test positive (Investigations) | 17 (17)
Headache (Nervous system disorders) | 35 (73)
Pyrexia (General disorders) | 37 (56)
Seasonal allergy (Immune system disorders) | 19 (24)
Vomiting (Gastrointestinal disorders) | 24 (33)
Cough (Respiratory, thoracic and mediastinal disorders) | 28 (52)
Upper respiratory tract infection (Infections and infestations) | 65 (164)
COVID-19 (Infections and infestations) | 40 (41)
Nasopharyngitis (Infections and infestations) | 40 (68)
Influenza (Infections and infestations) | 30 (36)
Pharyngitis streptococcal (Infections and infestations) | 27 (46)
Respiratory tract infection viral (Infections and infestations) | 22 (48)
Ear infection (Infections and infestations) | 18 (30)
Gastroenteritis (Infections and infestations) | 17 (22)
Bronchitis (Infections and infestations) | 15 (23)
Viral upper respiratory tract infection (Infections and infestations) | 15 (16)

LIMITATIONS AND CAVEATS:
The majority of enrollees were male, which is consistent with literature; Because GHD is a rare disease the study population size is modest.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-01-29): https://cdn.clinicaltrials.gov/large-docs/58/NCT03344458/Prot_000.pdf
  • Statistical Analysis Plan (2019-06-03): https://cdn.clinicaltrials.gov/large-docs/58/NCT03344458/SAP_002.pdf